CLINICAL TRIAL: NCT01563042
Title: An Exploratory First Time in Human (FTIH) Study Investigating the Pharmacokinetics (PK), Immunogenicity, Safety and Tolerability of GSK2434735 Administered as a Single Low Dose in Healthy Male Subjects
Brief Title: A Single Dose Pharmacokinetics (PK) Study of GSK2434735 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 114594
Record Dates: First submitted 2012-03-15; First posted 2012-03-26 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: immunogenicity; GSK2434735; pharmacokinetics (PK); PK; biospecific antibody
MeSH Terms: conditions — Asthma | interventions — Injections, Subcutaneous

ARMS (2):
- Cohort 1 GSK2434735 (Experimental): Cohort 1: Single intravenous administration of GSK2434735 and Pharmacokinetic (PK) and Immunogenicity assessments up to 42 days post dose.
  Interventions: Drug: Intravenous (IV) single dose
- Cohort 2 GSK2434735 (Experimental): Cohort 2: Single subcutaneous administration of GSK2434735 and Pharmacokinetic (PK) and Immunogenicity assessments up to 42 days post dose.
  Interventions: Drug: Subcutaneous (SC) single dose

INTERVENTIONS:
Drug: Intravenous (IV) single dose — GSK2434735 administered as a single intervenous dose at the beginning of the study
  Other Names: GSK2434735
  Arms: Cohort 1 GSK2434735
Drug: Subcutaneous (SC) single dose — GSK2434735 administered as a single subcutaneous dose at the beginning of the study
  Other Names: GSK2434735
  Arms: Cohort 2 GSK2434735

SUMMARY:
An exploratory First Time in Human (FTIH) study investigating the pharmacokinetics, immunogenicity, safety and tolerability of GSK2434735 administered as a single low dose in healthy male subjects

DETAILED DESCRIPTION:
Interleukin-13 (IL-13) and IL-4 are mediators in the pathogenesis of established asthmatic disease. GSK2434735 is a bispecific antibody to IL-13 and IL-4. The purpose of this open label, sequential cohort, exploratory First Time in Human (FTIH) study is to evaluate the pharmacokinetics (PK) profile of GSK2434735 after a single low intravenous or subcutaneous dose in healthy male volunteers, and to assess if the pharmacokinetics (PK) parameters can be scaled from monkey to man. In addition, the safety and tolerability will be monitored and the study will assess if antibodies are generated to GSK2434735.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 65 years of age
* Negative for pre-existing antibodies to GSK2434735.
* Body weight greater than and equal to 50 kg
* BMI 19 - 29.9 kg/m2.
* Lifelong non-smokers or ex-smokers of greater than 6 months

Exclusion Criteria:

* Clinically significant abnormalities.
* Current or past history of significant cardiac, respiratory, metabolic, renal, hepatic, neurological or gastrointestinal conditions.
* Current evidence or recent history of an infective illness.
* Vaccination within 3 weeks of screening
* History of severe allergic reactions, angio-oedema, anaphylaxis or immunodeficiency

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2012-05-23 (Actual); Study Completion 2012-05-23 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | 42 days
  Cmax, tmax, AUC, CL, t1/2

SECONDARY OUTCOMES:
Safety and tolerability of GSK2434735 as assessed by telemetry and change from baseline in 12-lead Electrocardiograms (ECG) | 42 days
  Change from baseline for PR, RR, QRS, QT, QTc measurements at Day 42
Safety and tolerability of GSK2434735 as assessed by change from baseline in blood pressure and heart rate | 42 days
  Change from baseline for systolic and diastolic blood pressure and heart rate measurements at 42 Days
Safety and tolerability of GSK2434735 as assessed by number of participants with adverse events | 42 days
  Clinically relevant changes from baseline in subject's disposition at Day 42
Change from baseline for Clinical laboratory assessments (hematology, chemistry and urinalysis | 42 days
  Changes from baseline values of hematologic , chemistry and urinary testing parameters at Day 42
Assessment of human anti-drug antibodies (ADA) in blood | 42 days
  Incidence of human anti-drug antibodies (ADA) at Day 42

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114594 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114594?search=study&search_terms=114594#rs
- Available data/document: Study Protocol: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114594 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register